CLINICAL TRIAL: NCT07088939
Title: Feasibility and Acceptability of a Self-guided Internet-delivered Dialectical Behavior Therapy Intervention for Adults With Mental Health Challenges
Brief Title: Feasibility and Acceptability of an E-learning Dialectical Behavior Therapy Skills Course
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Windsor (Other)
Responsible Party: Principal Investigator, Alexander Daros, Assistant Professor, University of Windsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-025
Record Dates: First submitted 2025-07-16; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Depression - Major Depressive Disorder; Anxiety; Depression; Stress; Mood Disorders
Keywords: dialectical behavior therapy; internet interventions; co-developed interventions; feasibility study; digital health
MeSH Terms: conditions — Anxiety Disorders; Depression; Mood Disorders | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered, self-guided dialectical behavior therapy (Experimental): Treatment arm
  Interventions: Behavioral: dialectical behavior therapy

INTERVENTIONS:
Behavioral: dialectical behavior therapy — This internet-delivered dialectical behavior therapy (iDBT) intervention consists of an e-learning course with 4 modules based on the 4 areas of skills training in dialectical behavior therapy: mindfulness, emotion regulation, distress tolerance, and interpersonal effectiveness. Participants can work through the modules at a self-guided pace to learn more than 30 specific skills using psychoeducational materials. The intervention incorporates psychoeducational elements of skills training with introductory videos, interactive quizzes, practice and homework suggestions, as well as quotes and videos from individuals with lived experience. In preliminary testing, it was estimated to take approximately 8-10 hours to complete all material.

SUMMARY:
Dialectical behavior therapy (DBT) is a comprehensive, third-wave psychological intervention designed for patients with complex and severe behavioral, emotional, and interpersonal dysfunction. DBT has since been adapted to shorter, briefer, "skills training" formats, which have been effective for a number of mild-to-moderate mental health conditions, including depression and anxiety. Moreover, internet-delivered formats of DBT (iDBT) have similarly started to build support for their effectiveness, although there are fewer studies on digital formats. One study found that over 12 weeks, iDBT was deemed acceptable (e.g., 50% of participants were still active after 4 weeks) and there were improvements in multiple symptom domains, such as depression, anxiety, suicidality, functional disability, as well as alcohol and substance dependence.

In the current study, the investigators will examine the feasibility, acceptability, and potential efficacy of a new iDBT intervention, packaged as an online e-learning skills course, with adult participants. The study is a pilot trial as iDBT has never been tested in this format through formal research. Thus, this pilot study aims to examine whether this course is usable, practical, and potentially useful to others in the future. The investigators will recruit up to 40 individuals with mild-to-moderate depression and anxiety for an 8-week study. Following a phone screen to determine eligibility, participants will complete a baseline session where they will provide consent, complete a brief interview and questionnaires, and register for the e-learning skills course. Over the course of 8 weeks, participants will be exposed to material adapted from a DBT manual in a self-guided manner. Participants will complete follow-up assessments at 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years old and up.
* Reside in Ontario.
* Fluent in English.
* Able to provide autonomous informed consent
* Reports at least mild depression and/or anxiety symptoms
* Not currently receiving any psychotherapy or psychosocial interventions.
* Have access to the internet

Exclusion Criteria:

* Practical (e.g., scheduling), acute psychiatric (e.g., suicidal ideation nearly every day, recent hospitalization for mental health reasons), or medical reasons (e.g., upcoming surgery, medical procedure, head injury).
* Not meeting one or more of the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability and Adherence Scale | 4 weeks and 8 weeks
  The Treatment Acceptability and Adherence Scale was used to assess ratings of perceived effectiveness, trustworthiness, and likelihood of adherence using a 7-point Likert scale from 1 (disagree strongly) to 7 (agree strongly). Items are summed to create a total score, with higher ratings indicating higher acceptability and adherence.
Intervention Usability Scale | 4 weeks and 8 weeks
  The Intervention Usability Scale is a 10-item measure to assess the ease of accessing and usability of the intervention. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). A total score is created by summing the items and higher ratings indicate higher usability of the intervention.

SECONDARY OUTCOMES:
Credibility and Expectancy Questionnaire | Baseline
  The Credibility and Expectancy Scale is used to assess whether participants had favorable opinions of the intervention and its potential effectiveness before starting treatment. In line with previous work, the first three items were used to evaluate credibility (using a 9-point Likert scale) whereas a single item (item 4) was used to evaluate expectancy of clinical improvement (using a 11-point Likert scale from 0% to 100%). The last two items are not scored.
Patient Health Questionnaire Depression Subscale | Baseline, 4 weeks, and 8 weeks
  The Patient Health Questionnaire Depression Subscale (PHQ-9) is a 9-item self-report measure used to assess depressive symptoms over the past two weeks. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). Items are summed to create a total score. Higher scores indicate greater depressive symptoms.
Generalized Anxiety Disorder 7 Questionnaire | Baseline, 4 weeks, and 8 weeks
  The Generalized Anxiety Disorder 7 Questionnaire (GAD7) is a 7-item self-report measure used to assess generalized anxiety symptoms over the past two weeks. Items are rated on a 4-point Likert scale from 0 (None at all) to 3 (Nearly Every Day). Items are summed to create a total score, with higher scores indicating greater symptoms.
World Health Organization Disability Assessment Schedule 2.0 Short Form | Baseline, 4 weeks, and 8 weeks
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) short form is a 12-item self-report measure assessing functional disability over the past month in several domains (cognition, mobility, self-care, getting along with others). Items are rated from 0 (none) to 4 (extreme or cannot do). Items are scored to create a total score. Higher scores indicate higher functional disability.
National Institute on Drug Abuse Assist for Alcohol and Substance Use | Baseline, 4 weeks, and 8 weeks
  The National Institute on Drug Abuse (NIDA) Assist is used to assess alcohol, smoking, and substance use involvement. This measure was used to assess alcohol, tobacco, cannabis, cocaine, amphetamine-type stimulants, inhalants, sedatives/sleeping pills, hallucinogens, and opioids. Each class of substance was rated for frequency over the past month using an ordinal scale: 0 (Never); 1 (Once or twice); 2 (3 or 4 times); 3 (5, 6, or 7 times); 4 (2 or 3 times a week); 5 (4 or 5 times a week); and 6 (Daily or almost daily). Ratings can be analyzed in terms of use at the binary level overall (indicating any substance used vs. no substances used) or at the class level (indicating one class was used vs. not used). Ratings can also be summed across substance classes with higher scores interpreted as greater frequencies of substance use.

OTHER OUTCOMES:
Difficulties in Emotion Regulation Scale, Short Form | Baseline, 4 weeks, and 8 weeks
  The Difficulties in Emotion Regulation Scale, Short Form (DERS-16; Kaufman et al., 2016) is a 16-item self-report measure, with excellent internal consistency, assessing emotion dysregulation based on a six-facet model first described by Gratz and Roemer (2004). Items are rated on a 5-point Likert scale from 1 (Almost Never) to 5 (Almost Always) and a total score is derived from summing the items (after reverse- scoring certain items). Higher scores reflect greater difficulties regulating emotions.
DBT Ways of Coping Checklist, Skills Subscale | Baseline, 4 weeks, and 8 weeks
  The DBT Ways of Coping Checklist (Neacsiu et al., 2010) is a 59-item self-report measure that assesses the frequency of maladaptive and adaptive skills used to manage difficult situations over the past month, with good internal consistency and test-retest reliability. In this study, the investigators only use the 38-item adaptive skills subscale, which includes skillful behaviors often learned in DBT without using DBT-specific language. Items were rated on a 4-point Likert scale from 0 (Never Used) to 3 (Regularly Used).
Mindful Awareness and Attention Scale (MAAS) | Baseline, 4 weeks, and 8 weeks
  The Mindful Awareness and Attention Scale (MAAS) is a 15-item measure of mindful attention and awareness, which is a primary target of DBT skills training. Items were rated on a 6-point Likert scale from 1 (Almost Never) to 6 (Almost Always). Higher scores reflect higher levels of dispositional mindfulness ability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Windsor, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No